CLINICAL TRIAL: NCT06363708
Title: Tislelizumab Combined With Chemotherapy as Neoadjuvant Treatment for Advanced Endometrial Cancer : A Prospective, Single-arm, Open-label Clinical Study
Brief Title: Tislelizumab in Combination With Chemotherapy as a Neoadjuvant Treatment for Advanced Endometrial Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024050
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Neoplasms
Keywords: Oncology; Endometrial Cancer; Tislelizumab
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — tislelizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab+Carboplatin+Paclitaxel (Experimental): Tislelizumab 200mg D1 +Carboplatin(AUC=5) D1+Paclitaxel(175 mg/m2 ) D1, every 3 weeks (21 days) is a treatment cycle
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg D1 ,Q3W
Drug: Paclitaxel — Paclitaxel(175 mg/m2 ) D1,Q3W
Drug: Carboplatin — Carboplatin(AUC=5) D1,Q3W

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of tislelizumab in combination with chemotherapy as a neoadjuvant treatment for advanced endometrial cancer.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm open-label study designed to enhance surgical R0 resection rate, reduce residual lesions, decrease distant metastasis and disease recurrence rates, and prolong the survival of patients with advanced endometrial cancer (stage III-IVb FIGO 2023) by neoadjuvant chemotherapy combined with tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signed informed consent form;
2. Age ≥18 years;
3. Eastern Cooperative Oncology Group performance status 0-1;
4. The International Federation of Gynecology and Obstetrics (FIGO 2023) stage III-IVb of endometrial cancer;
5. Has not received any systematic anti-tumor treatment for advanced diseases in the past;
6. Have measurable disease according to RECIST v1.1 criteria;
7. Patients must meet the following criteria for laboratory tests to ensure adequate organ function:

   * ANC ≥1,500/mm3, or ≥1.5×109/L
   * Platelet count≥75,000/mm3 or 75 x 109/L
   * Hemoglobin≥9 g/dL or ≥5.6 mmol/L
   * Glomerular filtration rate estimated（eGFR） according to the Chronic Kidney Disease Epidemiology Collaborative Group formula （CKD-EPI EQ6）was≥40 mL/ 1.73m2
   * Serum total bilirubin ≤ 1.5x upper limit of normal range（ULN）
   * Both AST and ALT were ≤3 x ULN
8. The expected lifespan exceeds 3 months.

Exclusion Criteria:

1. Received PD-1 target therapy other than tislelizumab or other antibody or drug therapy that specifically targets T-cell costimulation or checkpoint channels within 6 months before enrollment；
2. Has human immunodeficiency virus infection, active viral hepatitis, and active tuberculosis infection；
3. Active leptomeningeal disease or uncontrolled, untreated brain metastases resulting in elevated intracranial pressure;
4. Major surgical procedures had been performed within 4 weeks before consent was obtained；
5. Other conditions deemed by the investigator to be ineligible for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate (R0 %) | Up to approximately 24 months
  R0 resection rate is defined as the percentage of eligible patients that underwent a microscopically complete (or R0) resection. The resection is considered R0 if the inked margin is further than 1 mm distinct from any tumour cells.

SECONDARY OUTCOMES:
Pathological complete response rate (pCR%） | Up to approximately 24 months
  pCR is defined as the absence of invasive cells at microscopic examination of the primary tumor and lymph nodes at surgery. Any remaining in-situ lesions are permissible.
Objective Response Rate (ORR%) | Up to approximately 24 months
  ORR (either confirmed complete response [CR] or partial response [PR]) based on RECIST 1.1 will be determined in participants who have measurable disease at study entry.
Progression free survival (PFS) | Up to approximately 24 months
  PFS is defined as the time from the date of first dose to the earlier date of assessment of progression or death by any cause.
Recurrence free survival (RFS) | Up to approximately 24 months
  RFS is defined as the time from metastasectomy until progression by RECIST 1.1 or death from any cause.
Overall survival (OS) | Up to approximately 24 months
  OS is defined as time from first dose of study intervention to death from any cause.
Incidence and severity of adverse events as assessed by the NCI-CTCAE v5.0 | Up to approximately 24 months
  Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Hu, MD,PhD, Principal Investigator — Wuhan University
Locations (3):
- China (3):
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei maternal and child health care hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No